CLINICAL TRIAL: NCT01864083
Title: FACBC PET and PEM as a Staging Tool and Indicator of Therapeutic Response in Breast Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-177
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: FACBC PET/PEM; MR; 11-177
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- Local staging patients (Experimental): Breast MR and FACBC PET/PEM will be scheduled within one week of each other. Breast MR is a standard clinical examination and will be performed as standard.
  Interventions: Procedure: Positron Emission Tomography (PET); Drug: Fluorine-18 labeled 1-amino-3-fluorocyclobutane-1-carboxylic acid (FACBC); Procedure: Positron emission mammography (PEM) When available; Procedure: MR
- Neoadjuvant chemotherapy patients (Experimental): Baseline FACBC PET/PEM will be scheduled within 1 week of beginning neoadjuvant therapy. A repeat FACBC PET/PEM will be scheduled after the conclusion of neoadjuvant therapy, and before definitive surgical management.
  Interventions: Procedure: Positron Emission Tomography (PET); Drug: Fluorine-18 labeled 1-amino-3-fluorocyclobutane-1-carboxylic acid (FACBC); Procedure: Positron emission mammography (PEM) When available

INTERVENTIONS:
Procedure: Positron Emission Tomography (PET)
Drug: Fluorine-18 labeled 1-amino-3-fluorocyclobutane-1-carboxylic acid (FACBC)
Procedure: Positron emission mammography (PEM) When available
Procedure: MR
  Arms: Local staging patients

SUMMARY:
This study has been designed to help us determine if FACBC PET or PEM can accurately evaluate how far the breast cancer has spread in the breast. Also, to help determine if FACBC PET or PEM can accurately measure your response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for evaluation at MSKCC with biopsy proven primary IDC or ILC
* No prior therapy for IDC or ILC
* Clinical need for local disease staging with breast MR (Group A only)
* Clinical need for neoadjuvant chemotherapy (Group B only)
* Patients must provide written informed consent

Exclusion Criteria:

* Age <21 years
* Men
* Pregnancy or lactation
* Patients who have already started treatment for the current malignancy
* Patients who cannot undergo PET scanning (i.e. because of weight limits)
* Patients who are known to have contraindication for MRI (e.g. metal implants)
* Patients may only participate in group #1 or group #2, but not both

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
assess the diagnostic accuracy | 2 years
  Accuracy of standardized uptake values will be analyzed by receiver operating characteristic (ROC) curves. ROC curves will be constructed separately for FACBC PET, FACBC PEM and MR. The area under the curve will be used as a summary measure and compared using the standard nonparametric test [20]. We will also consider dichotomizing the uptake and present accuracy using sensitivity, specificity and predictive values. Dichotomized values will be compared using the McNemar test.
ability of FACBC PET and PEM to determine therapeutic response to neoadjuvant chemotherapy | 2 years
  Patients with locally advanced IDC or ILC, requiring neoadjuvant therapy prior to definitive surgery, will undergo FACBC PET and PEM both before chemotherapy and after. Following definitive breast surgery, pathologic specimens will be analyzed to determine if FACBC imaging can predict pathologic treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ulaner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Ulaner GA, Goldman DA, Corben A, Lyashchenko SK, Gonen M, Lewis JS, Dickler M. Prospective Clinical Trial of 18F-Fluciclovine PET/CT for Determining the Response to Neoadjuvant Therapy in Invasive Ductal and Invasive Lobular Breast Cancers. J Nucl Med. 2017 Jul;58(7):1037-1042. doi: 10.2967/jnumed.116.183335. Epub 2016 Nov 17. PMID 27856630
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/